CLINICAL TRIAL: NCT03318393
Title: Prospective Randomized Pilot Study Comparing Bivalirudin Versus Heparin in Neonatal and Pediatric Extracorporeal Membrane Oxygenation
Brief Title: Study Comparing Bivalirudin Versus Heparin in Neonatal and Pediatric ECMO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Lakshmi Raman, PROFESSOR, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 072017-045
Record Dates: First submitted 2017-10-04; First posted 2017-10-23 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-12

CONDITIONS: Extracorporeal Membrane Oxygenation Complication; Pediatric ALL; Anticoagulants
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — bivalirudin; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Unfractionated heparin group (Active Comparator): Patients randomized to this arm will undergo usual care using unfractionated heparin as the primary anticoagulant.
  Interventions: Drug: Unfractionated heparin
- Bivalirudin group (Experimental): Patients randomized to this arm will receive anticoagulation with bivalirudin
  Interventions: Drug: Bivalirudin

INTERVENTIONS:
Drug: Bivalirudin — Continuous infusion
  Arms: Bivalirudin group
Drug: Unfractionated heparin — Continuous infusion
  Arms: Unfractionated heparin group

SUMMARY:
The investigators will prospectively enroll 30 neonatal and pediatric ECMO patients at a single pediatric Level 1 trauma center. The patients will be randomized into two arms; one arm will receive unfractionated heparin and the other arm will receive bivalirudin. There will be 15 patients in each arm for a total of 30 patients.

Primary aim will be to compare the efficacy of bivalirudin to unfractionated heparin.

DETAILED DESCRIPTION:
The investigators will prospectively enroll 30 neonatal and pediatric ECMO patients at a single pediatric Level 1 trauma center. The patients will be randomized into two arms; one arm will receive unfractionated heparin and the other arm will receive bivalirudin. There will be 15 patients in each arm for a total of 30 patients.

The investigators hypothesize that neonatal and pediatric ECMO patients receiving bivalirudin will spend more time at goal anticoagulation and will experience less hemorrhagic and thrombotic complications when compared to patients receiving unfractionated heparin. Primary aim will be to compare the efficacy of bivalirudin to unfractionated heparin. The investigators secondary aim will be to define the incidence of hemorrhagic and thrombotic complications in patients receiving bivalirudin during ECMO.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 day to less than 18 years
* Cared for in the pediatric intensive care unit or pediatric cardiac intensive care unit
* receiving venovenous or venoarterial ECMO

Exclusion Criteria:

* Patients with known or suspected heparin induced thrombocytopenia prior to consent
* Patients with hepatic failure defined as coagulopathy with elevated transaminases more than three times normal values
* Patients with plan to decannulate from ECMO within 48 hours
* Known or suspected pregnant women
* Previous enrollment in this study
* Primary language spoken that is not English or Spanish

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2021-10-08 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ali McMichael, MD, Principal Investigator — UT Southwestern
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] McMichael A, Weller J, Li X, Hatton L, Zia A, Raman L. Prospective Randomized Pilot Study Comparing Bivalirudin Versus Heparin in Neonatal and Pediatric Extracorporeal Membrane Oxygenation. Pediatr Crit Care Med. 2025 Jan 1;26(1):e86-e94. doi: 10.1097/PCC.0000000000003642. Epub 2024 Nov 25. PMID 39585174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Unfractionated Heparin Group | Bivalirudin Group
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Unfractionated Heparin Group | Bivalirudin Group | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 14 | 16 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 7 | 5 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Spent at Goal Anticoagulation
Time Frame: through study completion, an average of 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Unfractionated Heparin Group | Bivalirudin Group
Number analyzed (Participants) | 14 | 16
percentage of time | 0.63 [0.5 to 0.82] | 0.49 [0.31 to 0.54]

2. Secondary Outcome: Number of Participants With One or More Major Bleeding Events
Description: Bleeding events will include drop in hemoglobin, surgical site bleeding, intracranial hemorrhage, fatal bleeding, extra surgical or unexpected surgical site bleeding
Time Frame: through study completion, an average of 1-2 weeks
Measure: Number; unit: participants
Arm/Group | Unfractionated Heparin Group | Bivalirudin Group
Number analyzed (Participants) | 14 | 16
participants | 7 | 7

3. Other Pre Specified Outcome: Number of Blood Products Transfused
Description: Will include fresh frozen plasma (FFP), packed red blood cells (pRBCs), platelets and cryoprecipitate
Time Frame: through study completion, an average of 1-2 weeks
Measure: Median (Inter-Quartile Range); unit: mls/kg/day
Arm/Group | Unfractionated Heparin Group | Bivalirudin Group
Number analyzed (Participants) | 14 | 16
mls/kg/day
  pRBCs | 12.2 [5.52 to 14.46] | 6.29 [2.49 to 8.41]
  Platelets | 13.58 [2.43 to 23.94] | 4.55 [0.55 to 11.51]
  FFP | 0.16 [0 to 2.84] | 1.15 [0.24 to 2.79]
  Cryoprecipitate | 0 [0 to 0.19] | 0.1 [0 to 1.14]

ADVERSE EVENTS:
Time Frame: From Baseline, daily until the end of study, an average of up to 0.1 year
Arm/Group | Unfractionated Heparin Group | Bivalirudin Group
All-Cause Mortality (participants affected / at risk) | 2/14 | 3/16
Serious Adverse Events (participants affected / at risk) | 7/14 | 7/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Unfractionated Heparin Group (N=14) | Bivalirudin Group (N=16)
Major bleeding event (Blood and lymphatic system disorders) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT03318393/Prot_SAP_000.pdf